CLINICAL TRIAL: NCT00022594
Title: Phase II Study Of NX 211 (Liposomal Lurtotecan) Given As An IV Bolus Injection On Days 1 and 8 Every 3 Weeks In Patients With Metastatic Or Loco-Regional Recurrent Squamous Cell Carcinoma Of The Head and Neck With Target Lesions Within Previously Irradiated Fields Or Outside Previously Irradiated Fields
Brief Title: Liposomal Lurtotecan in Treating Patients With Metastatic or Locally Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16008; EORTC-16008; GILEAD-110-10; OSI-EORTC-16008
Record Dates: First submitted 2001-08-10; First posted 2003-06-17 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

INTERVENTIONS:
Drug: liposomal lurtotecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of liposomal lurtotecan in treating patients who have metastatic or locally recurrent head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the therapeutic activity of lurtotecan liposome in patients with metastatic or loco-regionally recurrent squamous cell carcinoma of the head and neck.
* Determine the objective response, duration of response, and time to progression in patients treated with this drug.
* Determine the toxicity profile of this drug in these patients.
* Determine the possible pharmacokinetic/pharmacodynamic relationship of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to presence of a target lesion in a previously irradiated field (within vs outside).

Patients receive lurtotecan liposome IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 weeks.

PROJECTED ACCRUAL: A total of 38-72 patients (19-36 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck

  * Metastatic or loco-regionally recurrent disease
* No undifferentiated or non-keratinizing carcinomas including lymphoepitheliomas
* No tumors of the nasal or paranasal cavities or of the nasopharynx
* Measurable disease
* No clinical symptomatic evidence of brain or leptomeningeal metastases
* Ineligible for loco-regional treatment after chemotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* Transaminases no greater than 2.5 times ULN (5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 1.5 times ULN
* No uncontrolled hypercalcemia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after study
* No known hypersensitivity to systemic liposomal formulations or compounds chemically related to study drug
* No uncontrolled systemic disease or infection
* No psychological, familial, sociological, or geographical condition that would preclude study
* No other prior or concurrent malignancy except adequately treated cone-biopsied carcinoma in situ of the cervix or basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent anticancer biological therapy or immune response modifiers
* No concurrent prophylactic hematopoietic growth factors

Chemotherapy:

* See Disease Characteristics
* No prior chemotherapy for recurrent disease
* No prior therapy with camptothecin analogues
* At least 8 weeks since prior neoadjuvant or adjuvant chemotherapy
* No other concurrent anticancer cytotoxic therapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* At least 30 days since prior experimental drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-05; Primary Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Duffaud, MD, Study Chair — CHU de la Timone
Locations (20):
- Kaiser Franz Josef Hospital, Vienna (Wien), Austria
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- France (7):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer, Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - CHU de la Timone, Marseille
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - CHU Pitie-Salpetriere, Paris
  - Centre Henri Becquerel, Rouen
- Germany (2):
  - Universitats-Krankenhaus Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
- Italy (2):
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
- Netherlands (2):
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - University Medical Center Nijmegen, Nijmegen
- Instituto Portugues de Oncologia de Francisco Gentil-Centro de Lisboa, Lisbon, Portugal
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Switzerland (2):
  - Inselspital, Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- Royal Marsden NHS Trust, London, England, United Kingdom

REFERENCES:
- [Result] Duffaud F, Borner M, Chollet P, Vermorken JB, Bloch J, Degardin M, Rolland F, Dittrich C, Baron B, Lacombe D, Fumoleau P; EORTC-New Drug Development Group/New Drug Development Program. Phase II study of OSI-211 (liposomal lurtotecan) in patients with metastatic or loco-regional recurrent squamous cell carcinoma of the head and neck. An EORTC New Drug Development Group study. Eur J Cancer. 2004 Dec;40(18):2748-52. doi: 10.1016/j.ejca.2004.08.024. PMID 15571957